CLINICAL TRIAL: NCT01075698
Title: A Trial of Telmisartan Prevention of Cardiovascular Disease
Acronym: ATTEMPT-CVD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kumamoto University (Other)
Collaborators: Japan Foundation for Aging and Health (Other)
Responsible Party: Principal Investigator, Hirofumi Soejima, Associate Professor, MD, PhD, Kumamoto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H21-1
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: Type 2 Diabetes; Cerebrovascular disease; Coronary Artery Disease; Chronic Kidney Disease; Peripheral Artery Disease
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Cerebrovascular Disorders; Coronary Artery Disease; Renal Insufficiency, Chronic; Peripheral Arterial Disease | interventions — Standard of Care; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-ARB group (Active Comparator)
  Interventions: Drug: Non-ARB (standard therapy)
- ARB group (Active Comparator)
  Interventions: Drug: ARB (Telmisartan)

INTERVENTIONS:
Drug: Non-ARB (standard therapy) — Blood pressure lowering therapy except ARB
  Arms: Non-ARB group
Drug: ARB (Telmisartan) — Telmisartan 20-80 mg/day
  Arms: ARB group

SUMMARY:
The present research is conducted as a randomized, parallel-group, controlled, open study (using the PROBE method) to primarily verify the effects on various biomarkers in high-risk hypertensive patients treated with ARB (telmisartan, ARB group) as compared with those in patients receiving ordinary therapy (non-ARB group (ordinary therapy group)). In addition, onset of cardiovascular events and levels of markers that are associated with cardiovascular events are observed over time to examine the significance of each marker. The biomarkers will be obtained at the start of the study (at registration), after 6, 12, 24 and 36 months from the start of the study.

DETAILED DESCRIPTION:
Events are defined as follows; Cerebrovascular events: Stroke (cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, unknown type of stroke), transient ischemic attack Coronary events: Myocardial infarction, angina pectoris, asymptomatic myocardial ischemia Cardiac events: Myocardial infarction, angina pectoris, asymptomatic myocardial ischemia, heart failure Aortic/peripheral arterial events: Aortic aneurysm, aortic dissection, arteriosclerotic disease (aorta, carotid artery, renal artery, mesenteric artery, peripheral artery, etc.) Complications of diabetes: Diabetic nephropathy*, diabetic retinopathy*, diabetic neuropathy* Aggravation of renal function: Doubling of serum creatinine level, ESRD (initiation of dialysis, renal transplantation)

*Newly occurred or aggravated

The followings will be measured as biomarkers; urinary albumin creatinine rates (UACR), plasma brain natriuretic peptide (BNP), urinary 8-hydroxy-deoxy-guanosine (8-OHdG), serum adiponectin, serum high-molecular weight adiponectin, high sensitivity c-reactive protein (hsCRP), estimated glomerular filtration rate (eGFR)

ELIGIBILITY:
Inclusion Criteria: Patients who meet all of the criteria listed in [1] to [4] below and who have at least one cardiovascular risk listed in [1] to [5] below will be included in the study.

1. Outpatients
2. Age: ≥ 40 to < 80
3. Hypertension: Systolic blood pressure of ≥ 140 mmHg or diastolic blood pressure of ≥ 90 mmHg in the two latest measurements of casual blood pressure (in the sitting position) regardless of treated or untreated condition, or systolic blood pressure of < 140 mmHg and diastolic blood pressure of < 90 mmHg that require antihypertensive treatment.

   Assessment of hypertension: Blood pressure will be measured at least twice at an interval of 1 to 2 minutes. If the measured values obtained are substantially different, additional measurements will be performed and the average of two stable measurements will be used for assessment.
4. Patients who have given consent to participate in the present study.

Cardiovascular risks:

1. Diabetes mellitus; Type 2 diabetes mellitus
2. Kidney; Serum creatinine: 1.2 mg/dL - < 2.0 mg/dL for males, 1.0 mg/dL - < 2.0 mg/dL for females Proteinuria: qualitative value of ≥ +1 (quantitative value: proteinuria with the value of ≥ 0.3 g/g・Cr in casual urine when adjusted with urine creatinine) CKD stage 3 or higher (GFR < 60 mL/min/1.73 m2)
3. Heart; Previous myocardial infarction noted more than 6 months before obtaining the informed consent Diagnosis of angina pectoris Diagnosis of heart failure (NYHA I or II class) Diagnosis of left ventricular hypertrophy (left ventricular posterior wall of ≥ 12 mm evidenced by echocardiography performed prior to obtaining the informed consent, or Sv1+Rv5 of ≥ 35 mm noted as ECG finding) Diagnosis of transient or persisting atrial fibrillation
4. Brain; Previous cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage or transient cerebral ischemic attack noted more than 6 months before obtaining the informed consent
5. Peripheral arterial diseases; Previous lower-limb bypass surgery or angioplasty performed more than 6 months before obtaining the informed consent Ankle-brachial pressure index of < 0.9 or intermittent claudication

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

1. Type 1 diabetes mellitus
2. Severe renal disorders (serum creatinine of ≥ 2.0 mg/dL)
3. Myocardial infarction, percutaneous transluminal angioplasty and bypass surgery of coronary artery/ lower-limb blood vessel, cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage and transient cerebral ischemic attack noted within 6 months before initiation of the observation
4. Diagnosis of heart failure (NYHA III or IV class )
5. Virulent hypertension and secondary hypertension
6. Pregnant women
7. Clinically relevant allergic symptoms or past history of hypersensitivity to drugs / significant adverse drug reactions
8. Extremely poor bile secretion or serious liver disorders
9. Treatment-required malignant tumors
10. Patients who are judged by the physician in charge to be ineligible for the study for any other reasons

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1228 (Actual)
Dates: Start 2009-07; Primary Completion 2015-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The effects of ARB therapy and that of standard therapy except ARB on the biomarker levels (UACR and BNP) | for three years

SECONDARY OUTCOMES:
The effect of the two treatments on the incidence of events, and the relationship between the incidence of events and the biomarker levels (UACR, BNP, urine 8-hydroxy-2-deoxyguanosine, serum adiponectin, serum high-molecule adiponectin, eGFR) | for three years

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, Prof., MD, PhD, Study Chair — Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University; Shokei Kim-Mitsuyama, Prof., MD, PhD, Study Director — Department of Pharmacology and Molecular Therapeutics, Graduate School of Medical Sciences, Kumamoto University; Koichi Node, Prof, MD, PhD, Study Director — Department of Cardiovascular and Renal Medicine, Saga University Faculty of Medicine; Hirofumi Soejima, MD, PhD, Principal Investigator — Health Care Center / Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University; Osamu Yasuda, MD, PhD, Principal Investigator — Department of Cardiovascular Clinical and Translational Research, Kumamoto University Hospital
Locations (1):
- Department of Cardiovascular Clinical and Translational Research, Kumamoto University Hospital, Kumamoto, Japan

REFERENCES:
- [Background] Ogawa H, Soejima H, Matsui K, Kim-Mitsuyama S, Yasuda O, Node K, Yamamuro M, Yamamoto E, Kataoka K, Jinnouchi H, Sekigami T; ATTEMPT-CVD investigators. A trial of telmisartan prevention of cardiovascular diseases (ATTEMPT-CVD): Biomarker study. Eur J Prev Cardiol. 2016 Jun;23(9):913-21. doi: 10.1177/2047487315603221. Epub 2015 Aug 31. PMID 26324672
- [Derived] Kim-Mitsuyama S, Soejima H, Yasuda O, Node K, Jinnouchi H, Yamamoto E, Sekigami T, Ogawa H, Matsui K. Reduction in hsCRP levels is associated with decreased incidence of cardiovascular events in Japanese hypertensive women but not in men. Sci Rep. 2020 Oct 12;10(1):17040. doi: 10.1038/s41598-020-73905-4. PMID 33046765
- Available data/document: Study Protocol — https://prsinfo.clinicaltrials.gov/definitions.html